CLINICAL TRIAL: NCT07079137
Title: A Prospective Observational Study to Determine the Predictive Accuracy of Snakebite Severity Score (SSS) in Identifying Syndrome-Specific Core Outcome Parameters Amongst Envenomated Patients Presenting to the Emergency Department.
Acronym: SCOPE-Snake
Status: Not yet recruiting | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Dr Feba Susan Kurian, Junior Resident, Jubilee Mission Medical College and Research Institute
Other Study IDs: 67/25/IEC/JMMC&RI; U1111-1324-5906 (Other: World Health Organisation)
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Snake Bite
Keywords: snakebite; antivenom; snakebite severety score; modified snakebite severety score
MeSH Terms: conditions — Snake Bites | interventions — Health Records, Personal; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ● All patients 'clinically suspected snakebite' ● Presenting within 24 hours of the event ● Age ≥
  Interventions: Other: History, examination, bite documentation, SSS scoring,Baseline labs as per institutional protocol

INTERVENTIONS:
Other: History, examination, bite documentation, SSS scoring,Baseline labs as per institutional protocol — Following enrollment, an initial clinical assessment will be conducted in the Emergency Department (ED). This includes history taking, physical examination, documentation of bite characteristics, and calculation of the Snakebite Severity Score (SSS) at presentation. Baseline laboratory investigations will be performed as per institutional protocol.
  All participants will undergo serial clinical and laboratory monitoring as per institutional protocol. The development of syndrome-specific core outcomes, including neurotoxicity, haemotoxicity, coagulopathy, local tissue damage, acute kidney injury, and hypotension (Annexure) would be followed-up and evaluations will be conducted at the following time points:
  At presentation, Within 3 hours of ED admission, Within 6 hours of ED admission, Within 12 hours of ED admission

SUMMARY:
India reports ~58,000 snakebite deaths/year, over 50% of global mortality. Clinical outcomes of antivenom may vary due to regional venom differences, delayed access to care, ineffective use of existing polyvalent antivenom. There is a need for an India-specific severity assessment tool because it improves risk stratification & clinical decisions ,guides antivenom use, supports rural healthcare infrastructure, reduces morbidity, mortality, and financial burden.

Existing scoring systems lack validation for Indian envenomation patterns. Variability in venom (both inter- and intra-species) leads to inconsistent clinical outcomes.Misapplication of non-Indian tools may cause: Inaccurate severity grading, inappropriate antivenom use, poor patient outcomes.

PRIMARY OBJECTIVE:

● To determine the predictive accuracy of Snakebite Severity Score (SSS) done at the time of presentation in identifying syndrome specific core outcomes for snakebites.

SECONDARY OBJECTIVES:

* To evaluate the predictive accuracy of SSS in identifying patients at risk of mortality at 6 weeks
* To determine the predictive accuracy of modified Snakebite Severity Score (mSSS) done at the time of presentation in identifying syndrome specific core outcomes for snakebites

METHODOLOGY Study Duration: 18 months (Proposed)

* Setting: Emergency Dept, Jubilee Mission Medical College
* Sampling method :consecutive sampling
* Sample Size Calculation:

n = Z₍₁-α/₂)2 x SN (100-SN ) / l2 x P = 220

* Confidence Level: 95% (Z₍₁-α/₂₎ = 1.96)
* Expected Sensitivity: 97%
* Relative Allowable Error: 5% (l = 0.05)
* Proportion: Based on core outcome occurrence = 0.22
* Drop-out Rate Assumed: 20%
* minimum sample size = 264 Reference: Based on data from Dart et al."Validation of a Severity Score for the Assessment of Crotalid Snakebite,1999"

INCLUSION AND EXCLUSION CRITERIA

Inclusion Criteria:

* All patients 'clinically suspected snakebite'
* Presenting within 24 hours of the event
* Age ≥18 years
* Providing written informed consent

Exclusion Criteria

* Stings or bites other than snake
* All patients who received antivenom or blood products at another institute
* All patients with known hematological malignancies, coagulation disorders, chronic liver or renal failure
* All patients known to be on warfarin, heparin or any newer oral or injectable anticoagulants
* Individuals withdrawing a consent later on.

STUDY FLOW AND DATA MANAGEMENT

Study Flow:

Enrollment & Initial ED Assessment:

History, examination, bite documentation, SSS scoring Baseline labs as per institutional protocol

Monitoring & Follow-Up Timepoints:

T0: At presentation T+3h, +6h, +12h: Direct proforma, records review T+48h: Medical records Day 30 and Day 42 : Medical records & telephonic follow-up Outcomes Monitored: Neurotoxicity, haemotoxicity , coagulopathy, local damage, AKI, hypotension No interference with clinical care or treatment decisions.

DATA ANALYSIS PLAN:

Software: SPSS v29 Continuous variables are measured by using Mean+/-SD or median IQR Categorical variables are reported as frequencies and percentages. ROC curve analysis for SSS and mSSS. Logistic regression for mortality. Subgroup and domain-wise analysis.

ETHICAL CONSIDERATIONS:

Ethics approval to be obtained. Informed consent will be ensured. Data anonymized and securely stored. No interference with patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* All patients 'clinically suspected snakebite'
* Presenting within 24 hours of the event
* Age ≥18 years
* Providing written informed consent

Exclusion Criteria:

* Stings or bites other than snake
* All patients who received antivenom or blood products at another institute
* All patients with known hematological malignancies, coagulation disorders, chronic liver or renal failure
* All patients known to be on warfarin, heparin or any newer oral or injectable anticoagulants
* Individuals withdrawing a consent later on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients presenting to the Emergency Medicine Department of Jubilee Mission Medical College with clinically suspected snakebite envenomation will be screened for eligibility. Patients who meet the inclusion criteria and provide written informed consent will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine the sensitivity, specificity, negative predictive value (NPV), positive predictive value (PPV) and area under the curve (AUC) of the Snakebite Severity Score (SSS) recorded at the time of emergency department presentation | 2 years

SECONDARY OUTCOMES:
To evaluate the predictive accuracy of the SSS score at presentation in identifying patients who develop all-cause mortality within 6 weeks, using diagnostic performance metrics (AUC, sensitivity, specificity, PPV, NPV). | 2 years
To compare the predictive performance (AUC, sensitivity, specificity) of the Modified Snakebite Severity Score (mSSS) at presentation in detecting syndrome-specific core outcomes, over a 30-day follow-up period. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jubilee Medical Mission and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Undecided